CLINICAL TRIAL: NCT02979236
Title: Prospective, Observational, Italian Multi-center Registry of Self-aPposing cOronary Stent in Patients Presenting With ST-segment Elevation Myocardial InfarcTION: the iPOSITION Registry
Brief Title: Italian Multi-center Registry of Self-apposing Coronary Stent in Patients With STEMI
Acronym: iPOSITION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UOSD Emodinamica Diagnostica e Interventistica (Other)
Responsible Party: Principal Investigator, Livio Giuliani, MD PhD, UOSD Emodinamica Diagnostica e Interventistica
Other Study IDs: CH2016-01
Record Dates: First submitted 2016-11-24; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- STEMI treated with STENTYS Xposition S: Patients 18 years of age and older presenting with symptoms consistent with a ST-Elevation Myocardial Infarction (STEMI) lasting ≤12 hrs in duration, with ≥2 mm of ST-segment elevation in ≥2 contiguous leads, treated with primary stent implantation (Xposition S planned per operator's assessment).
  Interventions: Device: STENTYS Xposition S

INTERVENTIONS:
Device: STENTYS Xposition S

SUMMARY:
The aim of this registry is to collect clinical data on nitinol self-expanding STENTYS Xposition S™ in order to evaluate the efficacy and safety in patients presenting with ST segment elevation myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older presenting with symptoms consistent with a ST-Elevation Myocardial Infarction (STEMI) lasting ≤12 hrs in duration, with ≥2 mm of ST-segment elevation in ≥2 contiguous leads, treated with primary stent implantation (Xposition S planned per operator's assessment).

Exclusion Criteria:

* Cardiogenic shock
* Multiple lesions requiring stenting in the target vessel.
* Highly calcified lesions or excessive tortuosity at target lesion site.
* Intrastent pathology.
* Subject unable to take or comply with dual antiplatelet therapy as recommended per guidelines.
* Female subjects of childbearing potential known to be pregnant.
* Co-morbidities with life expectancy less than 1 year
* Patient unable to provide written informed consent.
* Known allergies to stent component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older presenting with symptoms consistent with a ST-Elevation Myocardial Infarction (STEMI) lasting ≤12 hrs in duration, with ≥2 mm of ST-segment elevation in ≥2 contiguous leads, treated with primary stent implantation (Xposition S planned per operator's assessment).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months post procedure
  target lesion failure will be assessed as the composite of cardiac death; recurrent Target Vessel-Related Myocardial Infarction (MI) and clinically driven Target Lesion Revascularization (TLR) by percutaneous or surgical methods (CABG).

SECONDARY OUTCOMES:
Procedural success without the occurrence of death and repeat ischemia-driven revascularization of the target lesion during the hospital stay | during the hospitalization, an average of 6 days
Target lesion failure at 30-day post-procedure | 30 day post procedure
Death from any cause | 12 months post procedure
Stent thrombosis rate at 30-day and 12-months after the procedure | 30 days post procedure and 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Livio Giuliani, MD PhD, Principal Investigator — UOSD Emodinamica Diagnostica e Interventistica
Locations (8):
- Italy (8):
  - Dipartimento cardiotoracico e vascolare - S.S Emodinamica Azienda Ospedaliera Nazionale SS Antonio e Biagio e Cesare Arrigo., Alessandria, Alessandria
  - UOC Cardiologia- UTIC Ospedale Civile "C. e G.Mazzoni", Ascoli Piceno, Ascoli Piceno
  - UOSD Emodinamica Diagnostica e Interventistica Ospedale SS Annunziata, Chieti, Chieti
  - UOC Terapia cardiologica intensiva ed interventistica Azienda Ospedaliera Universitaria G. Martino, Messina, Messina
  - UOC Cardiologia Emodinamica Ospedale San Salvatore - Centrale, Pesaro, Pesaro
  - UOC UTIC e Cardiologia Interventistica Ospedale S. Spirito, Pescara, Pescara
  - UOC Emodinamica Ospedale Umberto I, Syracuse, Siracusa
  - S.S. Emodinamica Ospedale San Giovanni Bosco, Torino, Torino

REFERENCES:
- [Background] Kim YS, Koo BK, Seo JB, Park KW, Suh JW, Lee HY, Park JS, Kang HJ, Cho YS, Chung WY, Chae IH, Choi DJ, Kim HS, Oh BH, Park YB. The incidence and predictors of postprocedural incomplete stent apposition after angiographically successful drug-eluting stent implantation. Catheter Cardiovasc Interv. 2009 Jul 1;74(1):58-63. doi: 10.1002/ccd.21961. PMID 19360868
- [Background] Gutierrez-Chico JL, Regar E, Nuesch E, Okamura T, Wykrzykowska J, di Mario C, Windecker S, van Es GA, Gobbens P, Juni P, Serruys PW. Delayed coverage in malapposed and side-branch struts with respect to well-apposed struts in drug-eluting stents: in vivo assessment with optical coherence tomography. Circulation. 2011 Aug 2;124(5):612-23. doi: 10.1161/CIRCULATIONAHA.110.014514. Epub 2011 Jul 18. PMID 21768536
- [Background] Foin N, Gutierrez-Chico JL, Nakatani S, Torii R, Bourantas CV, Sen S, Nijjer S, Petraco R, Kousera C, Ghione M, Onuma Y, Garcia-Garcia HM, Francis DP, Wong P, Di Mario C, Davies JE, Serruys PW. Incomplete stent apposition causes high shear flow disturbances and delay in neointimal coverage as a function of strut to wall detachment distance: implications for the management of incomplete stent apposition. Circ Cardiovasc Interv. 2014 Apr;7(2):180-9. doi: 10.1161/CIRCINTERVENTIONS.113.000931. Epub 2014 Mar 18. PMID 24642998
- [Background] Cook S, Eshtehardi P, Kalesan B, Raber L, Wenaweser P, Togni M, Moschovitis A, Vogel R, Seiler C, Eberli FR, Luscher T, Meier B, Juni P, Windecker S. Impact of incomplete stent apposition on long-term clinical outcome after drug-eluting stent implantation. Eur Heart J. 2012 Jun;33(11):1334-43. doi: 10.1093/eurheartj/ehr484. Epub 2012 Jan 26. PMID 22285579
- [Background] Nakano M, Yahagi K, Otsuka F, Sakakura K, Finn AV, Kutys R, Ladich E, Fowler DR, Joner M, Virmani R. Causes of early stent thrombosis in patients presenting with acute coronary syndrome: an ex vivo human autopsy study. J Am Coll Cardiol. 2014 Jun 17;63(23):2510-2520. doi: 10.1016/j.jacc.2014.02.607. Epub 2014 Apr 23. PMID 24768883
- [Background] Amoroso G, van Geuns RJ, Spaulding C, Manzo-Silberman S, Hauptmann KE, Spaargaren R, Garcia-Garcia HM, Serruys PW, Verheye S. Assessment of the safety and performance of the STENTYS self-expanding coronary stent in acute myocardial infarction: results from the APPOSITION I study. EuroIntervention. 2011 Aug;7(4):428-36. doi: 10.4244/EIJV7I4A71. PMID 21764660
- [Background] van Geuns RJ, Tamburino C, Fajadet J, Vrolix M, Witzenbichler B, Eeckhout E, Spaulding C, Reczuch K, La Manna A, Spaargaren R, Garcia-Garcia HM, Regar E, Capodanno D, Van Langenhove G, Verheye S. Self-expanding versus balloon-expandable stents in acute myocardial infarction: results from the APPOSITION II study: self-expanding stents in ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2012 Dec;5(12):1209-19. doi: 10.1016/j.jcin.2012.08.016. PMID 23257368
- [Background] Koch KT, Grundeken MJ, Vos NS, IJsselmuiden AJ, van Geuns RJ, Wessely R, Dengler T, La Manna A, Silvain J, Montalescot G, Spaargaren R, Tijssen JG, Amoroso G. One-year clinical outcomes of the STENTYS Self-Apposing coronary stent in patients presenting with ST-segment elevation myocardial infarction: results from the APPOSITION III registry. EuroIntervention. 2015 Jul;11(3):264-71. doi: 10.4244/EIJY15M02_08. PMID 25692610
- [Background] van Geuns RJ, Yetgin T, La Manna A, Tamburino C, Souteyrand G, Motreff P, Koch KT, Vrolix M, IJsselmuiden A, Amoroso G, Berland J, Montalescot G, Teiger E, Christiansen EH, Spaargaren R, Wijns W. STENTYS Self-Apposing sirolimus-eluting stent in ST-segment elevation myocardial infarction: results from the randomised APPOSITION IV trial. EuroIntervention. 2016 Feb;11(11):e1267-74. doi: 10.4244/EIJV11I11A248. PMID 26865444
- [Background] Grundeken MJ, Lu H, Mehran R, Cutlip DE, Leon MB, Yeung A, Koch KT, Montalescot G, van Geuns RJ, Spaargaren R, Buchbinder M. APPOSITION V: STENTYS coronary stent system clinical trial in subjects with ST-segment elevation myocardial infarction--rationale and design. Am Heart J. 2014 Nov;168(5):652-60. doi: 10.1016/j.ahj.2014.07.011. Epub 2014 Jul 24. PMID 25440792
- [Background] Sianos G, Papafaklis MI, Serruys PW. Angiographic thrombus burden classification in patients with ST-segment elevation myocardial infarction treated with percutaneous coronary intervention. J Invasive Cardiol. 2010 Oct;22(10 Suppl B):6B-14B. PMID 20947930